CLINICAL TRIAL: NCT05604703
Title: Comparison of Two Different Periodontal Disease Classifications At the Patient Level
Brief Title: Comparison of Different Periodontal Classifications
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Berceste Guler, Principal Investigator, Kutahya Health Sciences University
Other Study IDs: 2021/02-06
Record Dates: First submitted 2022-10-30; First posted 2022-11-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-08

CONDITIONS: Periodontal Diseases
Keywords: 2018 new periodontal classification; periodontal diseases; Armitage periodontal classification
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Periodontal classification — 300 patients will be classified according to 1999 armitage and 2018 new periodontal classification and compared.

SUMMARY:
Due to some deficiencies in the classification defined by Armitage in 1999, a new periodontal classification was published in 2018. New periodontitis A staging and grading system was used for classification. Staging depends largely on the severity of the disease, while grading is based on the rate of disease progression to the past. It provides additional information on a risk-based analysis and assessment of risk.The aim of this study is to reveal the differences between the old periodontal classification and the new periodontal disease classification published in 2018. Periodontitis in the literature review. The two classifications were compared in patients. However, a study on gingival recession not done. Anamnesis, routine periodontal indices, routine radiographs of 300 patients, first of all According to the 1999 Periodontal Disease Classification, after it will be classified according to the New Periodontal Disease Classification developed in 2018. Thus, two different Periodontal Disease Classifications, old and new, comparison will be made.

DETAILED DESCRIPTION:
In the 1999 periodontal disease classification, the diagnosis of chronic and aggressive periodontitis was subdivided into localized and generalized. Chronic periodontitis is an inflammatory disease of supporting tissues followed by pocket formation, gingival recession, periodontal ligament, alveolar bone and attachment loss. Aggressive periodontitis is characterized by rapid periodontal attachment loss and alveolar bone loss in which the patient is systemically healthy, inherited, and the presence of Aggregatibacter Actynomyecetemcomitans in diseased areas.

Due to some deficiencies in the classification defined by Armitage1 in 1999, the need for a new periodontal classification emerged in 2018. These shortcomings are;

1. There is no specific evidence of pathophysiology that differentiates cases into "aggressive" or "chronic" periodontitis or guides different types of treatment.

2 There is little evidence that aggressive and chronic periodontitis are different diseases. However, there is evidence that multiple factors and their interactions influence clinically observable disease outcomes (phenotypes) at the individual level.

3. On a population basis, average rates of periodontitis progression are consistent across all populations observed worldwide. However, there is evidence that certain segments of the population exhibit different levels of disease progression.

4. A classification system based solely on disease severity; It fails to capture important dimensions of an individual's disease, such as the complexity of treatment approaches and the risk factors that affect disease outcomes.

For this reason, a new periodontal classification was published in 2018.2 The staging and grading system was used in the new periodontitis classification. Staging largely depends on the severity of the disease at presentation and the complexity of disease management. Staging consists of four categories (stages 1 to 4) and is determined by considering various variables such as clinical attachment loss, amount and percentage of bone loss, probing depth, presence and extent of angular bone defects, and furcation involvement, tooth mobility, and tooth loss. Grading, on the other hand, provides additional information about a historical analysis of the rate of disease progression, further progression of the biological characteristics of the disease, including an assessment of risk, the expected poor outcome of treatment, and the assessment of the risk that the disease or its treatment may adversely affect the patient's overall health.

The Miller3 classification used for gingival recession is based on the position of the marginal gingiva3. In the new classification, the classification of gingival recessions has also been updated. Recent case definitions for the treatment of gingival recession are based on interproximal loss of clinical attachment and also include assessment of exposed root and enamel-cementum margin. A new classification of gingival recession, including clinical parameters, has added the gingival phenotype as well as the features of the exposed root surface. The term periodontal biotype has been replaced by periodontal phenotype.

The aim of this study is to reveal the differences between the old periodontal classification and the new periodontal disease classification published in 2018. In the literature4 review, two classifications were compared in patients with periodontitis. However, no research has been conducted on gingival recessions. Our aim is to compare the cases of gingivitis, periodontitis and gingival recession according to two different classifications.

Anamnesis of all patients who applied to KSBU Faculty of Dentistry, Department of Periodontology, routine periodontal indices and routine radiographs are taken. This index of all patients and Radiographs are used in the diagnosis and classification of periodontal diseases. disease Classification is important for guiding treatment. For this reason, all patients Classification is routinely done. This study was conducted for periodontal surgery after pre-examination.

300 patients with indications will be included. Routine periodontal surgery from these patients, like other patients, indexes and radiographs will be taken. Comparison of the two classifications these indexes and radiographs will be made through By examining the indices and radiographs taken from the patients, the patients were first It will be classified according to the old Periodontal Disease Classification. The same indexes and New Classification of Periodontal Diseases developed in 2018 using radiographs will be determined. Thus, two different Periodontal Disease Classifications, old and new, comparison will be made.

Routine indexes used:

* Plaque index (Löe & Silness) and gingival index (Silness & Löe) are obtained by measuring 4 regions of a tooth (mesial, distal, buccal and lingual) with Williams periodontal probe.
* Attachment loss: The distance between a tooth and the free gingiva based on the enamel-cementum boundary is measured using a Williams periodontal probe.
* Bleeding index on probing (Ainamo & Bay): In this index, probing is performed by gently walking around the pocket. As a result of probing, the evaluation is made by looking at the presence or absence of bleeding in the gingiva. A positive value is given if bleeding occurs within 10-15 seconds after probing in the mesial, distal, buccal and lingual parts of all teeth. The ratio of the bleeding area to the examined area is expressed as %.
* Keratinized gingival width: It is the distance from the free gingival margin to the mucogingival junction line.
* Pocket depth: It is the vertical distance between the base of the periodontal sulcus and the gingival margin with a standard periodontal probe measured.
* Peri-implant pocket depth: The vertical distance between the base of the peri-implant sulcus and the gingival margin
* Presence of diabetes: It is questioned whether the patient has diabetes or not.
* Smoking: Whether the patient smokes or not, and if so, the amount is questioned.
* Gingival recession: It is the apical migration of the marginal gingiva from the enamel-cementum junction. It can be evaluated clinically by measuring the distance in mm between the enamel-cementum junction (MSB) and the gingival gingival margin.
* Chronic Periodontitis: It is the presence of interdental clinical attachment loss in more than 2 non-adjacent teeth, or a pocket depth ≥3 mm in the buccal or oral region in more than 2 teeth, in addition to clinical attachment loss ≥3 mm.
* Localized Aggressive Periodontitis: Attachment loss is observed in the proximal regions of the first molar and incisors. Loss of proximal attachment is observed in at least 2 permanent teeth, one of which is the first molar. More than two teeth should be unaffected except for the molars and incisors.
* Generalized Aggressive Periodontitis: 1. At least 3 more teeth are affected except molars and incisors.

Routine radiographs used:

* Panoramic Radiography: X-ray imaging that allows the evaluation of the lower and upper jaws and all teeth on the same film. It is routinely taken from all patients for the diagnosis of periodontal disease.
* Periapical Radiography: It is an X-ray imaging that provides a more detailed examination of one or several adjacent teeth. It is routinely taken from all patients for the diagnosis of periodontal disease.

Periodontal disease classification of patients is made by determining the number of missing teeth, type of bone destruction and the tooth with the highest bone loss on panoramic and periapical radiographs, and calculating the bone loss/age ratio of this tooth in millimeters.

* Panoramic Radiography: X-ray imaging that allows the evaluation of the lower and upper jaws and all teeth on the same film. It is routinely taken from all patients for the diagnosis of periodontal disease.
* Periapical Radiography: It is an X-ray imaging that provides a more detailed examination of one or several adjacent teeth. It is routinely taken from all patients for the diagnosis of periodontal disease.

Periodontal disease classification of patients is made by determining the number of missing teeth, type of bone destruction and the tooth with the highest bone loss on panoramic and periapical radiographs, and calculating the bone loss/age ratio of this tooth in millimeters.

Statistical analysis method: Descriptive assessments will be made. SPSS software will be used. Chi-square test will be applied for analysis.

ELIGIBILITY:
Inclusion Criteria:

* be over 18 years old
* Patients with recorded periodontal indices and radiographs
* Patients without disease affecting bone metabolism

Exclusion Criteria:

* Mentally retarded patients
* Pregnant and breastfeeding patients
* Patients receiving radiotherapy
* Patients who do not use drugs that impair bone metabolism such as bisphosphonates

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Apply to Kütahya University of Health Sciences, Faculty of Dentistry, Department of Periodontology.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Number of aggressıve or chronic periodontitis patients according to 1999 armitage periodontal classification | T0=baseline
  The age and systemic diseases of the patient are learned and the pocket depth, alveolar bone and attachment loss are measured and classified as localized or generalized with aggressive or chronic periodontitis.
New periodontal classifıcatıon stage | T0=baseline
  Number of patients according to Staging depends on the severity of the disease; clinical attachment loss, amount and percentage of bone loss, probing depth, angular the presence and extent of bone defects and furcation involvement, tooth mobility, and tooth loss. determined by considering the variables.
New periodontal classifıcatıon grade | T0=baseline
  Number of patients according to Grading is based on the rate of disease progression. It reflects an analysis based on diabetes and varies depending on the HbA1c value if the patient has diabetes, the number of cigarettes smoked, and the bone loss/age ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Berceste Güler, Study Director — Kütahya Health Sciences University
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Department of Periodontology, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data can be shared if the principal investigator is contacted.
Supporting Information: Study Protocol, CSR
Time Frame: After the research paper is published.
Access Criteria: The IPD will be shared if the principal investigator is contacted.

REFERENCES:
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370
- [Background] Caton JG, Armitage G, Berglundh T, Chapple ILC, Jepsen S, Kornman KS, Mealey BL, Papapanou PN, Sanz M, Tonetti MS. A new classification scheme for periodontal and peri-implant diseases and conditions - Introduction and key changes from the 1999 classification. J Clin Periodontol. 2018 Jun;45 Suppl 20:S1-S8. doi: 10.1111/jcpe.12935. PMID 29926489
- [Background] Miller PD Jr. A classification of marginal tissue recession. Int J Periodontics Restorative Dent. 1985;5(2):8-13. No abstract available. PMID 3858267
- [Background] Graetz C, Mann L, Krois J, Salzer S, Kahl M, Springer C, Schwendicke F. Comparison of periodontitis patients' classification in the 2018 versus 1999 classification. J Clin Periodontol. 2019 Sep;46(9):908-917. doi: 10.1111/jcpe.13157. Epub 2019 Jun 28. PMID 31152600
- [Background] Guttiganur N, Aspalli S, Sanikop MV, Desai A, Gaddale R, Devanoorkar A. Classification systems for gingival recession and suggestion of a new classification system. Indian J Dent Res. 2018 Mar-Apr;29(2):233-237. doi: 10.4103/ijdr.IJDR_207_17. PMID 29652020